CLINICAL TRIAL: NCT05266222
Title: Respiratory Virus Sampling and Repository
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000707; 000707-I
Record Dates: First submitted 2022-03-03; First posted 2022-03-04 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09-09

CONDITIONS: Influenza; COVID-19
Keywords: Influenza; Flu; COVID; Coronavirus; Immunity; Natural History
MeSH Terms: conditions — Influenza, Human; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with respiratory infection: Persons with suspected or documented respiratory infection

SUMMARY:
Background:

Respiratory viruses, like the flu or COVID-19, cause significant illness and death worldwide. Researchers want to collect samples from people with respiratory virus infections. The samples in this natural history study will be used in future research.

Objective:

To obtain samples from people with respiratory viruses to learn more about respiratory virus infections and the immune responses against them.

Eligibility:

People aged 3 and older who have or are suspected to have a respiratory virus infection.

Design:

Participants will be screened with a medical record review.

Participants will give blood samples. Data from their medical records will be collected.

Participants will give nose samples. A soft plastic strip will be put into each nostril for a minute. They may also give nose, mouth (back of the throat), or saliva samples using swabs.

Participants may receive kits by mail to collect nose and blood samples at home. They will use soft plastic strips to collect nose samples. To collect blood, they will prick their finger and dab a few drops of blood on four plastic tips.

If a participant is in the hospital, air samples may be collected in their room.

Participation will last for up to 2 years. After 2 years, participants may be asked for their consent again to give new samples and new medical data.

DETAILED DESCRIPTION:
Study Description:

Retrospective and prospective samples from participants will be obtained to isolate respiratory viruses for use in laboratory assays, animal experiments, development of challenge virus, and development of vaccines. Samples will also be obtained to study respiratory virus-associated systemic and mucosal immunity and virus characteristics.

Objectives:

Primary Objective:

To isolate human respiratory virus specimens and maintain them in a repository for future use in laboratory assays, animal experiments, development of challenge viruses, and development of vaccines, described in a separate protocol.

Study Population: 1-200 (for each virus species/strain) adult and child participants aged 3 years and above with suspected or documented respiratory infection for a maximum of 20000 participants total. The total number of subjects enrolled will depend on the prevalence of infection with each virus/strain and on the geographic distribution of infections.

Description of Sites/Facilities Enrolling Participants:

NIH Clinical Center (CC).

Study Duration: 10 years

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Aged 3 years or older.
2. Documented or suspected infection with a respiratory virus.
3. Stated willingness to comply with all study procedures for the duration of the study.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any condition that, in the opinion of the investigator, would compromise the safety of the study participant or staff, or would prevent proper conduct of the study.

Non-English Speaking Participants: This study will enroll non-English speaking participants.

For non-English speaking participants, the study will be explained to the participant/family through an interpreter, in the presence of the study team, in the language understood by the participant/family. The short form in the language understood by the participant/family will be signed by the participant/family or LAR and the interpreter, and the consent will be signed by the consenting provider and the interpreter.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons with suspected or documented respiratory infection
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To isolate human respiratory virus specimens | 10 years
  To isolate human respiratory virus specimens and maintain them in a repository for future use in laboratory assays, animal experiments, development of challenge viruses, and development of vaccines, described in a separate protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NIH Building 33 (NIAID), Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No
We are not working with any outside collaborators that require this information

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000707-I.html